CLINICAL TRIAL: NCT00203606
Title: Effectiveness of Pegylated Interferon Plus Ribavirin in the Treatment of Active and Past Intravenous Drug Users Infected With Hepatitis C
Brief Title: Pegylated Interferon Plus Ribavirin in the Treatment of Active and Past Intravenous Drug Users Infected With Hepatitis C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Roche Pharma AG (Industry)
Responsible Party: Robert Hilsden, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21995
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Hepatitis c
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Treatment (Experimental): Active Treatment with Pegylated Interferon Alfa 2a (Pegasys, Roche) and ribavirin
  Interventions: Drug: pegylated interferon alfa-2a ( Roche) and ribavirin
- Observation (No Intervention): Observation with no active treatment for Hepatitis C. Observation period is based on standard treatment duration based on genotype of Hepatitis C. Active treatment offered to participants at conclusion of observation. (Protocol Amendment #1, October 30, 2001. Ethics approval Jan 19, 2004).

INTERVENTIONS:
Drug: pegylated interferon alfa-2a ( Roche) and ribavirin — pegylated interferon alfa-2a ( Roche) and ribavirin
  Arms: Active Treatment

SUMMARY:
Hepatitis C infects as many as 300,000 Canadians. Up to 25% of those infected will develop cirrhosis and be at risk for liver failure and liver cancer. Cirrhosis caused by hepatitis C is the most common reason for liver transplantation in Canada. The largest group of infected people are those who use injectable street drugs. However, people who continue to use drugs are routinely excluded from scientific studies testing new treatments for Hepatitis C and are generally recommended not to receive available treatments. Although several reasons are given to justify excluding these people from treatment, little scientific evidence is available to support it. We plan to examine how successful treatment with the current standard treatment of pegylated interferon and ribavirin is in those who continue to use injection drugs. We will compare the results of treatment of 70 active drug users to results of published clinical trials (this is a change from initial plan to compare to treatment results of 70 local) reformed drug users). Our goal is to determine whether reasonable success rates can be achieved in active drug users that would then further justify their routine treatment.

DETAILED DESCRIPTION:
We plan to examine how successful treatment with the current standard treatment of pegylated interferon and ribavirin is in those who continue to use injection drugs. Our goal is to determine whether reasonable success rates can be achieved in active drug users that would then further justify their routine treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women age 18 to 75 years.
2. Chronic hepatitis C infection based on a history of positive anti-HCV antibody and/or HCV RNA at least 6 months prior to study entry.
3. Positive HCV-RNA by Roche Amplicor HCV test at screening
4. Serum ALT > 1.5 times upper limit of normal
5. Active or past use of injection drugs or crack cocaine by self-report. Active use is defined as injection drug use at least 1/month and within 3 months of the date of randomization. Past use is defined as no injection drug use or crack cocaine use within the past 5 years.
6. Compensated liver disease
7. Negative urine or blood pregnancy tests (for women of childbearing potential) documented within 24-hours prior to first dose of study drug.
8. All fertile males and females must use effective contraception during treatment and during the 6 months after treatment end if sexually active (This will be provided free of charge to active IDUs).

Exclusion Criteria:

1. Presence of clinically evident ascites requiring active diuretic therapy, history of or therapy for hepatic encephalopathy, or history of variceal bleeding within the last two years.
2. Platelet count < 60,000/mm3
3. Serum ALT level > 10 times upper limit of normal
4. Serum creatinine level > 1.5 times the upper limit of normal (Deleted February 27, 2007, Protocol Amendment #4, Ethics approval March 28, 2007)
5. Hematology outside of specified limits: neutrophil count < 1000/mm3, hemoglobin < 10 g/L in males and < 9 g/L in females

7. Unstable or uncontrolled thyroid disease 8. Treatment with interferon- and/or ribavirin within the previous 12 months 9. Presence of clinically significant cryoglobulinemia vasculitis (e.g. skin rash, arthritis, or renal insufficiency due to cryoglobulinemia) 10. Presence or history of autoimmune hepatitis, alpha-1-anti-trypsin deficiency, genetic hemochromatosis, Wilson disease, drug- or toxin-induced liver disease, alcohol-related liver disease, primary biliary cirrhosis, or sclerosing cholangitis.

11. Chronic hepatitis B infection or positive HbsAg at screening 12. Known history of HIV infection or positive HIV antibody test by Western Blot.

13. A disease known to cause significant alteration in immunologic function, including hematological malignancy or autoimmune disorder.

14. Concurrent therapy with immunosuppressive drugs or cytotoxic agents, such as prednisone, cyclosporine, azathioprine or chemotherapeutic agents.

15. History of unstable or deteriorating cardiac, pulmonary or renal disease. 16. Preexisting (within last two years) or active psychiatric condition including severe untreated depression, major psychoses, suicidal ideation or suicidal attempts.

17. Severe or poorly controlled diabetes mellitus 18. Any serious or chronic disease that may affect the assessment of safety or efficacy parameters.

19. Patients who have had a liver transplant 20. Patients infected with HCV genotypes 4, 5 or 6 (< 1% of infected current/past IDUs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2004-01; Primary Completion 2009-01 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Sustained viral response | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Hilsden, MD PhD, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - Pender Clinic, Vancouver, British Columbia